CLINICAL TRIAL: NCT03366441
Title: Effective Methods for Reactivating Inactive Blood Donors: a Stratified Randomized Controlled Study
Brief Title: Reactivation of Inactive Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Principal Investigator, OUYANG Jian, Principal Investigator, Guangzhou Blood Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Guangzhou Blood Center
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Blood Donor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telephone group (Experimental): The telephone group received telephone calls. All non-response and refusing donors were included for further follow-up. Donors who answered the phone call and agreed to be interviewed were asked the reasons why they had stopped donating according to a pre-designed questionnaire. All of the responsed donors were re-recruited by altruistic appeal.
  Interventions: Other: Telephone call
- SMS group (Experimental): The SMS intervention group received the following text message:"Dear donors, Thank you for your donation through which your love brought hope to those helpless patients and your donated blood reignited the fire in their lives. If you can, please consider donating blood again to save a life. Thank you again for your support!" . All donors either receiving or not receiving the message were included for further follow-up.
  Interventions: Other: SMS
- Control group (No Intervention): No intervention will be giving to this group.

INTERVENTIONS:
Other: Telephone call — From 20 October to 10 November 2016, telephone calls were given to the donors in the phone call group
  Arms: Telephone group
Other: SMS — Text messages were sent to an equal number of donors in the SMS group
  Arms: SMS group

SUMMARY:
Blood donor retention is a critical strategy to ensure the safety and sufficiency of clinical blood supply. An effective strategy can prevent donors from lapsing and eventually becoming inactive.

ELIGIBILITY:
Inclusion Criteria:

* Donated blood at least once between Januanry 1 to September 30 2016, and the blood test result is qualified.

Exclusion Criteria:

* Having donated again before intervened.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11880 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Blood donation rate | 1 year
  Number of blood donors donate blood again divided by the number of participants in every group after intervened.

SECONDARY OUTCOMES:
Self-deferral reasons of not donating | 1 day
  The reasons of not donating again in the telephone group.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China